CLINICAL TRIAL: NCT03182673
Title: A Phase I, Open Label, Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SHR7390 Combined With SHR-1210 and SHR3162 in Patients With Advanced Solid Tumors
Brief Title: The Study of SHR7390 in Combination With SHR-1210 and SHR3162 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR7390-I-102-AST
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumor
Keywords: advanced solid tumor; Protein Kinase MEK inhibitor (MEKi); Programmed Death 1(PD-1); Safety; Pharmacokinetics; PARP inhibitor
MeSH Terms: interventions — camrelizumab; fluzoparib; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Intervention Model Description: SHR7390,SHR-1210 and SHR3162
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR7390, SHR-1210 and SHR3162 (Experimental): Total 60-100 subjects with advanced solid tumors
  In the two-drug combination therapy,subjects were received single oral doses of SHR7390，then accepted two drug combination therapy, SHR7390 is administered multiple daily oral doses of SHR7390 for 28 days for a treatment cycle. At the same time, SHR-1210 was given intravenously per 2 weeks at the 200mg fixed dose.
  In the second study part, subjects accepted three drug combination therapy, SHR7390 is administered orally for 21 days and discontinued for 7 days in a 28-day treatment cycle,SHR3162 was administered orally twice a day for 28 days at a fixed dose of 100 mg. At the same time, SHR-1210 was given intravenously per 2 weeks at the 200mg fixed dose
  Interventions: Drug: SHR7390; Biological: SHR-1210; Drug: SHR3162

INTERVENTIONS:
Drug: SHR7390 — SHR7390 is provided as white, film-coated,immediate release tablets containing SHR7390 at dosage strengths of 0.125 mg,0.5 mg and 2mg. Multiple tablets of SHR7390 will be administered orally to achieve targeted doses of SHR7390: 0.125 mg-4 mg. Tablets will be administered once daily or for 21 days and discontinued for 7 days with 240 ml water after 2 hours of the meal.
  Other Names: MEKi
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 immunoglobulin G4 (IgG4) monoclonal antibody. SHR-1210 is provided as the lyophilized powder,200 mg/vial.SHR-1210 was given with 200mg fixed dose intravenously per 2 weeks at the D1 and D15.Intravenous infusion over 30 min
  Other Names: PD-1
Drug: SHR3162 — SHR3162 is provided as capsules containing SHR3162 at dosage strengths of 10mg,40mg and 100mg. The capsule of SHR3162 will be orally administered with 240ml water twice a day to achieve targeted doses of SHR3162 and the interval of SHR3162 capsules taken twice a day is about 12 hours.
  Other Names: parp inhibitor

SUMMARY:
The study consists of the two parts, the first one is SHR7390 combined with SHR-1210, the second one is SHR7390 combined with SHR-1210 and SHR3162. Two parts of the study are separately to assess the safety and tolerability, to define dose limiting toxicity（DLT) and maximum tolerated dose (MTD),to evaluate the pharmacokinetics ,to assess the antitumor activity in patients with advanced solid tumors preliminarily and to recommend reasonable dosage regimen of SHR7390 for the follow-up clinical trial.

DETAILED DESCRIPTION:
This is a phase I, open-label,two parts,dose escalation/expansion clinical study.The safety,tolerance,PK and preliminary efficacy of two-drug combination and three-drug combination were evaluated respectively in the patients with advanced solid tumors that have no any targeted agents as the standard therapies.

In the first study part, subjects receiving a single dose of SHR7390 (Run-in) are observed in 7-10 days, then accepted two drug combination therapy, SHR7390 is administered once daily orally for 28 days for a treatment cycle. At the same time, SHR-1210 was given intravenously per 2 weeks at the fixed dose of 200mg.

In the second study part, subjects accepted three drug combination therapy, SHR7390 is administered orally for 21 days and discontinued for 7 days in a 28-day treatment cycle,SHR3162 was administered orally twice a day for 28 days at a fixed dose of 100 mg. At the same time, SHR-1210 was given intravenously per 2 weeks at the fixed dose of 200mg.

Dose limiting toxicities (DLT) in the first study part will be assessed during the Run-in and first cycle of treatment. the dose escalation is designed by Accelerated Titration Designs during initial accelerated phase. when the significant toxicity or DLT is observed in the Run-in and first cycle of treatment,the accelerated titration trial terminates and subsequent dose escalations are become a conventional design of 3+3 patients. If one adverse event （AE） meets dose limiting toxicity (DLT) criteria at a given dose, 3 additional patients will be enrolled in this dose cohort. If 2 DLTs are determined at a given dose level, the previous dose will be designated as the MTD.

Based on preliminary determination of RP2D and sufficient safety data in the first part of the study, the second part of three-drug combination will be carried out. the preset dose of SHR7390 includes RP2D initially determined in the first part of the study and its previous low dose level (for example, RP2D is 0.5 mg/d, while the former low dose is 0.25 mg/d). Dose escalation is a conventional design of 3+3 patients.

Additional patients will be enrolled for pharmacokinetic (PK) evaluations at different dose levels based on preliminary safety and tolerability.Each dose level can expand at least 12 subjects , of which 9-12 subjects are PK subjects. Multiple blood samples at designated time points will be collected for PK evaluations (more than 12 subjects are determined by SMC).

The safety, tolerability and AEs will be closely monitored throughout the study duration. The preliminary effectiveness and clinical benefits of two-drug combination and three-drug combination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

The study is open to all males and females who meet the following inclusion criteria at screening and baseline to participate in the study.

To be included to participate in this study each patient must:

1. 18-70 years of age, both male and female;
2. The invalid standard treatment or non standard and effective treatment in patients with advanced solid tumors diagnosed by pathology;

（1) in the phase of dose escalation , the subjects with RAS or BRAF mutation status and microsatellite stability （MSS）are not restricted.

（2）in the phase of dose expansion，the subjects with RAS or BRAF mutations and microsatellite stability (MSS) are included necessarily.

（3) the subjects included in the phase of dose expansion must have at least one measurable target lesion with RECIST V 1.1.

(4) If they in the phase of dose expansion are unable to provide the results of previous RAS/BRAF mutation and microsatellite stability,subjects must provide previous cancer tissues（paraffin blocks or pathological 8-10 white sections）, or fresh biopsy specimens.

3. The Eastern Cooperative Oncology Group （ECOG） General status (performance status, PS) of 0-1;

4. The expected lifetime ≥ 3 months;

5. The organ function must meet the following requirements:

1. Adequate bone marrow reserve: including neutrophil absolute count,platelets and hemoglobin;
2. Liver: serum albumin ≥ 2.8 g/dl; bilirubin≤1.5 upper limit of normal value (ULN), Alanine aminotransferase（ALT）and aspartate aminotransferase（AST）≤ 2.5 upper limit of normal value (ULN),if there is liver metastasis, the ALT or AST≤5xULN;
3. Kidneys: creatinine clearance ≥ 50 mL/min (Cockcroft-Gault of the standard formula）；
4. Heart: left ventricular ejection fraction ≥ 50%; normal Electrocardiograph (ECG) and corrected QT interval（QTc）;male QTc<450ms，female QTc<470ms

6. The lesion of the patients caused by other treatments has been restored(≤1 grade，except alopecia and other adverse events that the investigators judged to be tolerable）。The time interval between previous treatment and the first use of study drugs：nitrosourea or mitomycin> 6 weeks; cytotoxic drugs, monoclonal antibodies, radiotherapy or surgery> 4 weeks; TKI targeted drugs> 2 weeks;endocrine therapy> 1 week；

7. A agreement to use a highly effective, non-hormonal form of contraception is required for women of childbearing potential and men with partners of childbearing potential, who were not sterilized surgically, for duration of the study treatment and after the last dose of study treatment; For female patients of child bearing potential,who was not sterilized surgically,the serum human chorionic gonadotropin （HCG） pregnancy test must be the negative

8. Voluntary ability to follow the procedures of clinical study. Written informed consent is provided by signing the informed consent form.

Exclusion Criteria:

1. Previous treatment with any other tumor immune checkpoint inhibitors within 2 months before the first use of study drugs；previous treatment with other MEK inhibitors or PARP inhibitors (the previous treatment of PARP inhibitors is only excluded in the second part of the study).
2. Use of other investigational anti-cancer drugs or the termination of the investigational drugs within the last four weeks.
3. The subjects had active autoimmune diseases, a history of immunodeficiency disease and autoimmune diseases, or a history of disease or syndrome with systemic steroid hormones or immunosuppressive drugs(such as asthma, idiopathic pulmonary fibrosis, institutional pneumonia, bronchiolitis obliterans, and drug pneumonia,idiopathic pneumonia or interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis,hyperthyroidism, hypothyroidism, but not limited to these diseases or syndromes），or other acquired (HIV) and congenital immunodeficiency diseases, or a history of organ transplantation (including allogeneic bone marrow transplantation).
4. Known severe hypersensitivity or other hypersensitivity to chimeric or humanized antibodies or fusion proteins; known to be allergic or hypersensitive to components of SHR-1210，SHR7390 or SHR3162.
5. The subjects were known to have tumor metastases of central nervous system or meningeal metastases, or a history of primary tumors of CNS.
6. Presence of a factor that influences the oral drug (such as inability to swallow) or presence of active gastrointestinal disease or other diseases that will interfere significantly with the absorption, distribution, metabolism, or excretion of drug.
7. History of the retinopathy or the sensory retinal detachment. As assessed by ophthalmologist, presence of the risk factors of study treatment that may cause retinal vein thrombosis/occlusion (RVO), central serous chorioretinopathy (CSCR),or neovascular and macular degeneration.
8. The intraocular pressure > 21mmHg or glaucoma was diagnosed within 4 weeks
9. The evidence of severe or uncontrollable pleural effusion, peritoneal effusion or pericardial effusion. The clinical treatment is required, such as periodic drainage.
10. The evidence of severe or uncontrolled systemic diseases (e.g. chronic lung, liver, kidney, or heart diseases).
11. Unstable angina pectoris or new angina pectoris within recent three months.Presence of arrhythmia, myocardial ischemia with long-term drug treatment.III-IV stage heart failure as defined by the New York Heart Association (NYHA). Presence of acute myocardial infarction events and congestive heart failure within the first six months before screening.
12. Medical treatment for an acute stage of infection or active TB.
13. Hepatitis B virus（HBV) or hepatitis C virus (HCV) infection stage with abnormal liver function.
14. Pregnant or lactating women or intending to become pregnant during the study period.
15. Living attenuated vaccines within one months of the initial use of the drug, or a living attenuated vaccine is expected during the study period.
16. A history of neurological or psychiatric disorders, and a history of psychotropic substance or drug abuse.
17. According to the judgement of the investigators, presence of serious hazards to the safety of the subjects, the concomitant diseases confusing to analyze the study data or influencing to complete this study (such as severe hypertension, diabetes, thyroid disease, etc.),or any other situation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose-Limiting Toxicity(DLT) | up to 24 months
  A DLT is considered at AE related to study drug unless there is a clear, well-documented, alternative explanation for the toxicity. Severity of AEs are graded according to the NCI CTCAE 4.03 for the study, the occurrence of the following drug related AEs during the single dose and the first cycle(35-38 days,two-drug combination) or the first cycle (28 days, three-drug combination) will be considered a DLT by the investigator and SMC.
  MTD is the highest dose of SHR7390 in subjects with DLT less than 33.3% during the DLT observation in the dose escalation of two-drug combination.

SECONDARY OUTCOMES:
The assessment of Treatment-related Adverse Events | Up to 24 months
  Assessment of the incidence and severity of treatment-related AEs in all subjects who received at least 1 dose of SHR7390,SHR-1210 and SHR3162.
Time to peak (Tmax) of plasma concentration | up to 24 months
  Pharmacokinetics profile of SHR7390:Time to peak (Tmax) of plasma concentration
Maximum plasma concentration (Cmax) | up to 24 months
  Pharmacokinetics profile of SHR7390: Maximum plasma concentration (Cmax)
Halflife (T1/2) | up to 24 months
  Pharmacokinetics profile of SHR7390: Halflife (T1/2)
Clearance/ bioavailability (CL/F) | up to 24 months
  Pharmacokinetics profile of SHR7390: Clearance/ bioavailability (CL/F)
apparent volume of distribution/bioavailability (Vd/F) | up to 24 months
  Pharmacokinetics profile of SHR7390: apparent volume of distribution/bioavailability (Vd/F)
Area under curve (AUC) | up to 24 months
  Pharmacokinetics profile of SHR7390: Area under curve (AUC)
Accumulation index (Rac) | up to 24 months
  Pharmacokinetics profile of SHR7390: Accumulation index (Rac)
blood concentration of SHR7390 | up to 24 months
  Pharmacokinetics profile of SHR7390:blood concentration
plasma concentration of SHR7390 | up to 24 months
  Pharmacokinetics profile of SHR7390:plasma concentration
plasma concentration of SHR3162 | up to 24 months
  Pharmacokinetics profile of SHR3162: plasma concentration
serum concentration of SHR-1210 | up to 24 months
  Pharmacokinetics profile of SHR-1210: serum concentration
Efficacy Assessments | up to 24 months
  Subjects will be assessed using RECIST v1.1. The primary aim is to demonstrate clinically meaningful improvement in ORR.
The identification of the recommended Phase 2 dose (RP2D) of SHR7390 in subjects with advanced solid tumors | up to 24 months
  When the dose escalation is accomplished, RP2D will be identified by the characterization of safety.

CONTACTS AND LOCATIONS:
Overall Officials: RuiHua Xu, MD, PhD, Principal Investigator — The Cancer Center,Sun Yat-sen University
Locations (1):
- The Cancer Center,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No